CLINICAL TRIAL: NCT00001677
Title: Methotrexate Alone Versus Combination of Methotrexate and Subcutaneous Fludarabine for Severe Rheumatoid Arthritis: Safety, Tolerance and Efficacy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980117; 98-AR-0117
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Arthritis, Rheumatoid; Synovitis
Keywords: Immunosuppression; Lymphocytes; Magnetic Resonance; Synovial Biopsy; Synovitis; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Synovitis | interventions — Methotrexate; fludarabine

INTERVENTIONS:
Drug: Methotrexate
Drug: Fludarabine

SUMMARY:
The safety profile and efficacy of combination therapy will be evaluated using methotrexate (MTX) and the nucleoside analog fludarabine in 40 patients with severe refractory rheumatoid arthritis. The patients enrolled will be those who have experienced inadequate disease control with MTX alone or in combination with other immunosuppressive drugs such as sulfasalazine (SSZ), cyclosporin A (CsA), or hydroxychloroquine (HCQ). In this randomized, double-blind, placebo controlled trial, patients will be maintained on oral MTX at 17.5 mg/week to which either placebo or subcutaneous fludarabine at 30 mg/m(2) daily for three consecutive days per month will be added for four months. The fludarabine (or placebo) treatment period will be followed by two months of follow-up, at which time patients will be evaluated for response. Patients will be monitored for adverse effects/tolerability, disease activity, and changes in synovial volume as measured by magnetic resonance imaging (MRI). Additionally synovial biopsies will be obtained before and after treatment for investigation of infiltrating cell numbers and phenotypes, cytokine profiles, Th1 versus Th2 responses, and angiogenesis.

DETAILED DESCRIPTION:
The safety profile and efficacy of combination therapy will be evaluated using methotrexate (MTX) and the nucleoside analog fludarabine in 40 patients with severe refractory rheumatoid arthritis. The patients enrolled will be those who have experienced inadequate disease control with MTX alone or in combination with other immunosuppressive drugs such as sulfasalazine (SSZ), cyclosporin A (CsA), or hydroxychloroquine (HCQ). In this randomized, double-blind, placebo controlled trial, patients will be maintained on oral MTX at 17.5 mg/week to which either placebo or subcutaneous fludarabine at 30 mg/m(2) daily for three consecutive days per month will be added for four months. The fludarabine (or placebo) treatment period will be followed by two months of follow-up, at which time patients will be evaluated for response. Patients will be monitored for adverse effects/tolerability, disease activity, and changes in synovial volume as measured by magnetic resonance imaging (MRI). Additionally synovial biopsies will be obtained before and after treatment for investigation of infiltrating cell numbers and phenotypes, cytokine profiles, Th1 versus Th2 responses, and angiogenesis.

ELIGIBILITY:
Ability to provide informed consent to all aspects of the study after full information is provided.

Age equal to or older than 18.

A diagnosis of Rheumatoid Arthritis (RA) of more than 6 months as defined by the revised American College of Rheumatology criteria.

Active RA defined as: 6 or more swollen joints;

6 or more tender joints;

ESR greater than 28 mm/hr (or CRP greater than 0.8) or morning stiffness greater than 45 minutes.

Incomplete response (defined as persistently active disease as described above) to treatment with at least one of the following regimens for over 3 months:

MTX alone (greater than or equal to 17.5 mg/week);

MTX (greater than or equal to 17.5 mg/week) plus HCQ (greater than or equal to 200 mg/day);

MTX (greater than or equal to 17.5 mg/week) plus SSZ (greater than or equal to 1 gm/d);

MTX (greater than or equal to 17.5 mg/week) plus CsA (1-3 mg/kg/day);

MTX (greater than or equal to 17.5 mg/week) plus SSZ (greater than 1 gm/day) plus HCQ (greater than or equal to 200 mg/day);

No requirement of corticosteroids in doses equivalent to over 10 mg/d prednisone nor other immunosuppressive agents required for the control of extraarticular manifestations at the time of study entry.

No active acute or chronic infections requiring antibiotic therapy, serious viral infections (such as hepatitis, herpes zoster, or HIV), or serious fungal infections. Patients with a positive PPD who have not received INH or other antituberculous therapy will be excluded.

No pregnant women, nursing mothers, or patients of childbearing age not practicing birth control.

No preexisting malignancy other than basal cell carcinoma.

No history of stroke, seizure disorder, or chronic neurologic disease.

No unstable coronary artery disease, cardiomyopathy, conduction heart block greater than first degree, or a dysrhythmia requiring therapy.

No confounding medical illness that in the judgment of the investigators would pose added risk for study participants (e.g., chronic hepatic, renal, or pulmonary disease or bone marrow hypoplasia).

No presence of seronegative spondyloarthropathy, systemic lupus erythematosus, systemic sclerosis, inflammatory myopathy, systemic vasculitis, psoriasis, or inflammatory bowel disease.

No serum creatinine greater than 2.0 mg/dL on at least 2 different occasions which is sustained for at least 1 month.

No hematocrit less than 28% (or hemoglobin less than 9.0 mg/dL), or platelet count less than 100,000, or white blood count less than 3,500/dL.

No patients with active lung disease, patients with a chronic and progressive lung disease, or patients with a chronic but stable lung disease with pulmonary function tests of less than 70% of predicted (DLCO less than 60%).

No patients with hypogammaglobulinemia (IgG count less than 300).

No patients treated with alkylating agents for over 1 year at any time or treated with a purine nucleoside analog at any time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1998-06; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Priebe T, Platsoucas CD, Seki H, Fox FE, Nelson JA. Purine nucleoside modulation of functions of human lymphocytes. Cell Immunol. 1990 Sep;129(2):321-8. doi: 10.1016/0008-8749(90)90208-9. PMID 1696525
- [Background] Davis JC Jr, Fessler BJ, Tassiulas IO, McInnes IB, Yarboro CH, Pillemer S, Wilder R, Fleisher TA, Klippel JH, Boumpas DT. High dose versus low dose fludarabine in the treatment of patients with severe refractory rheumatoid arthritis. J Rheumatol. 1998 Sep;25(9):1694-704. PMID 9733448